CLINICAL TRIAL: NCT02824718
Title: A Randomized Crossover TrIal to Compare Recombinant Human rhPTH(1-34) to the ASsociation Alfacalcidol/Hydrochlorothiazide in the Treatment of Severe Primary Hypoparathyroidism
Brief Title: Recombinant Human rhPTH(1-34) VS Association Alfacalcidol/Hydrochlorothiazide in Severe Primary Hypoparathyroidism
Acronym: ACTICAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P150911; PHRC-15-549 (Other Grant/Funding Number: Ministry of health, France); 2016-000500-29 (EudraCT Number)
Record Dates: First submitted 2016-07-01; First posted 2016-07-07 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Autosomal Dominant Hypocalcemia OR Primary Hypoparathyroidism Related to Other Cause But Complicated by Hypercalciuria Under Treatment
Keywords: Hypoparathyroidism; PTH(1-34); Thiazides; Hypercalciuria; Calcium sensing receptor
MeSH Terms: conditions — Hypoparathyroidism; Hypercalciuria | interventions — Teriparatide; Thiazides; Hydrochlorothiazide; Sodium Channel Blockers; Amiloride; alfacalcidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rh PTH(1-34) (Experimental): 40 µg/day rhPTH(1-34) (teriparatide or FORSTEO® 20 µg twice daily) over 7 to 8 weeks (52±3 days).
  Interventions: Drug: Teriparatide
- Thiazide + potassium sparing diuretic (Active Comparator): hydrochlorothiazide 25 mg/day (ESIDREX®) + amiloride 5 mg/day (MODAMIDE®) + 0.5 µg/day alfacalcidol (ALFACALCIDOL®) over 7 to 8 weeks (52±3 days).
  Interventions: Drug: Thiazide; Drug: Potassium sparing diuretic; Drug: Alfacalcidol

INTERVENTIONS:
Drug: Teriparatide — human recombinant parathormone
  Other Names: FORSTEO
  Arms: rh PTH(1-34)
Drug: Thiazide — Diuretic
  Other Names: ESIDREX
  Arms: Thiazide + potassium sparing diuretic
Drug: Potassium sparing diuretic — Diuretic
  Other Names: MODAMIDE
  Arms: Thiazide + potassium sparing diuretic
Drug: Alfacalcidol — Belongs to the class of vitamin D and analogues
  Other Names: UN-ALFA
  Arms: Thiazide + potassium sparing diuretic

SUMMARY:
Hypoparathyroidism is a rare condition in which the parathyroid glands fail to produce sufficient amount of parathyroid hormone or the parathyroid hormone produced lacks biologic activity. The most common cause of hypoparathyroidism is damage to or removal of the parathyroid glands due to neck surgery for another condition. Occurrence of hypercalciuria under treatment is a frequent concern in primary hypoparathyroidism, limiting correction of hypocalcemia.

Hypoparathyroidism can also be caused by an autoimmune process. In rare cases, hypoparathyroidism may occur as a genetic disorder inherited as an autosomal recessive, autosomal dominant or X-linked recessive trait. The autosomal dominant hypocalcemia (ADH) is mainly caused by heterozygous activating mutations in the CASR gene encoding CaSR). As other severe presentation of primary hypothyroidism, ADH is characterized by the increased risk to develop hypercalciuria and nephrolithiasis. The purpose of the study is to compare two therapeutic approaches in severe hypoparathyroidism in order to limit the risk of nephrocalcinosis and renal failure when attempting to correct hypocalcemia: rhPTH(1-34) vs association of active vitamin D and hydrochlorothiazide. The European Society of Endocrinology Clinical has indeed recently published guidelines for the treatment of chronic hypoparathyroidism in adults. These guidelines suggest considering treatment with a thiazide diuretic In a patient with hypercalciuria and replacement therapy with PTH in patients who do not stably and safely maintain their serum and urinary calcium in the target range.

DETAILED DESCRIPTION:
The design consists in a five-periods, two-treatments, open-label, randomized, crossover study with blind end-point evaluation.

Patients will come for an inclusion visit and will receive treatment with 0.5 µg/day alfacalcidol for 4 weeks (28±3 days, run-in). They will be instructed to maintain dietary calcium intakes (1 g/day) for the duration of the study and will be supplemented throughout the study with native vitamin D in order to maintain the concentration of 25OH vitamin D ≥ 40 ng/L. Magnesium supplementation (100 mg/day) will be maintained throughout the study.

At inclusion, patients will be randomly assigned to receive at the end of run-in period, in cross-over either an association hydrochlorothiazide 25 mg/day (ESIDREX®) + amiloride 5 mg/day (MODAMIDE®) + 0.5 µg/day alfacalcidol (ALFACALCIDOL®) or 40 µg/day rhPTH(1-34) (teriparatide or FORSTEO® 20 µg twice daily) over 7 to 8 weeks (52±3 days).

After a washout period of 28±3 days under 0.5 µg alfacalcidol /day, the patients will follow the second period of treatment. The study will end with a final period of 28±3 days under 0.5 µg alfacalcidol /day. Patients will ambulatory monitor serum calcium, sodium, potassium, and creatinine levels at days 15 of run in and run out periods and at day 7 and day 28 of each treatment period.

ELIGIBILITY:
Inclusion criteria :

* Patients aged from 18 to 80 years, of both sexes
* Patient with primary hypoparathyroidism related to a genetically proven ADH OR primary hypoparathyroidism related to other cause but complicated by hypercalciuria under treatment
* Affiliated to a French health insurance system, and who have consented to the study.

Exclusion criteria :

* Pregnant and breastfeeding women;
* Women of childbearing age without contraception;
* For men aged from 18 to 20 years, presence of cartilage of growth on X-ray of left knee;
* Anuria;
* Kidney failure with plasmatic creatinine >125 mmol/l and urea >10 mmol/l;
* Long QT interval : QTc > 450 ms (men) or 470 ms (women);
* Hepatic failure;
* Metabolic bone diseases (Paget's disease of bone) other than primary osteoporosis or glucocorticoid-induced osteoporosis;
* Association to other potassium sparing diuretics;
* Hypokalemia (<3.5 mmol/l) without diuretic therapy;
* Hyperkalemia (>5.5 mmol/l);
* Hyponatremia (<135 mmol/l) without diuretic therapy;
* Hypercalcemia (>2.6 mmol/l);
* Severe hypomagnesemia (≤ 0.5 mmol/l);
* Vitamin D deficiency (25OH vit D < 20 ng/mL);
* Unexplained increase in alkaline phosphatase (>2N);
* Intolerance to sulfamide;
* Intolerance to amiloride or other component of the drug;
* Hypersensitivity to any active substance or excipient of one of the experimental drugs;
* Gluten intolerance;
* Bone break history within the three previous months;
* History of radiotherapy of the skeleton;
* History of bone cancer or metastasis.
* Personnal or familial (first degree relatives) of skin cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Plasma calcium concentration | two months of treatment
  Mean of two measures at 30-min interval of Ionized serum calcium concentration

SECONDARY OUTCOMES:
Ambulatory calcium concentration | days 7 an 28 of treatment by rhPTH(1-34) and association alfacalcidol/hydrochlorothiazide and at day 14 of non-treatment periods (run in, wash out, run out).
  Ambulatory measurement of serum calcium level
Calciuria | Inclusion, weeks 4 (end of the run-in period), 7-8 (end of the first treatment period), 11-12 (end of the wash-out period), 18-20 (end of the second treatment period), 202 (end of the wash-out period)
  24h-urinary calcium excretion (expressed as mmol/24h and mmol/mmol creatinine)
Plasma calcium x phosphate product | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
Blood pressure | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
Serum sodium level | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
Serum potassium level | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
Estimated GFR using MDRD formula | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
Serum renin level | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
Serum aldosterone level | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
24h-urinary sodium excretion | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
24h-urinary potassium excretion | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
24h-urinary aldosterone excretion | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
Serum 25 OH vitamin D level | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
Serum 1,25(OH)2 vitamin D level | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
Serum magnesium level | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
24h-urinary magnesium excretion | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Tolerance of thiazides and amiloride
Calcium/citrate ratio measured on spot urines | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Assessment of stone formation risk
Calcium/creatinine ratios measured on spot urines | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Assessment of stone formation risk
Crystalluria | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Assessment of stone formation risk
Alkaline phosphatase level | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Evaluation of the impact of rhPTH(1-34) on bone
Number of episodes of cramps | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Other tolerance
Number of episodes of paresthesia | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Other tolerance
Number of episodes of tetany | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Other tolerance
Number of episodes of seizure | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Other tolerance
SF36 self-administered questionnaire | Inclusion, days 28 (end of the run-in period), 80 (end of the first treatment period), 108 (end of the wash-out period), 160 (end of the second treatment period), 202 (end of the wash-out period)
  Evaluation of the impact on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Anne Blanchard, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Agnes Linglart, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP Hopital Europeen Georges Pompidou, Paris, France